CLINICAL TRIAL: NCT00927888
Title: The Effect of Preemptive Sphenopalatine Ganglion Block on Anesthetic Requirements, Postoperative Pain and Functional Patient Outcomes After Functional Endoscopic Sinus Surgery
Brief Title: Postoperative Pain and Functional Patient Outcomes After Functional Endoscopic Sinus Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: Hospira, now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Principal Investigator, David R. Drover, Professor, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SU-05072009-2478
Record Dates: First submitted 2009-06-23; First posted 2009-06-25 (Estimated); Results first posted 2015-03-04 (Estimated); Last update posted 2016-05-19 (Estimated); Status verified 2016-04

CONDITIONS: Pain, Postoperative
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 - Bupivacaine Block (Active Comparator): 3 ml of 0.25% Bupivacaine with Epi 1:100,000 (A block)
  Interventions: Drug: Bupivacaine Block
- 2 - Placebo (Placebo Comparator): Normal saline with Epi 1:100,000 (B block)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Bupivacaine Block — Bupivacaine local anesthesia block prior to start of FESS procedure.
  Other Names: Local Block
  Arms: 1 - Bupivacaine Block
Drug: Placebo — placebo is identical in appearance in comparison to active drug.
  Other Names: Placebo saline injection
  Arms: 2 - Placebo

SUMMARY:
The aim of the study is to quantify postoperative pain after functional endoscopic sinus surgery (FESS) and investigate whether preemptive analgesia may positively impact intraoperative anesthetic management, decrease patient postoperative pain and discomfort, and improve patient functional outcomes.

DETAILED DESCRIPTION:
The sphenopalatine ganglion block (SPGB) with local anesthetic is used to treat facial pain and headache of various etiologies and has been widely used during functional endoscopic sinus surgery (FESS). The purpose of this study was to investigate whether preemptive SPGB may positively impact postoperative pain and functional outcomes after FESS.

A prospective, double-blind randomized placebo-controlled study was performed. 60 patients (18 to 70 yrs), undergoing general anesthesia for bilateral FESS, were randomly assigned to receive SPGB with either 2 ml 0.25% bupivacaine with epinephrine 1:100,000 (BP, treatment group) or normal saline (NS, control group). SPGB was performed preemptively 10 min before the start of surgery. Pre- and post operative (day#0, day#7, day#30) visual analogue pain scale, SNOT-20, CT & Endoscopic scores were compared between the two groups.

ELIGIBILITY:
Inclusion Criteria:

1. The study subjects will be 18-70 year old.
2. The subjects will be American Society of Anesthesiology physical status I and II patients.
3. Patients with chronic rhinosinusitis, presenting for bilateral functional endoscopic sinus surgery.
4. The subjects should understand informed consent and study instructions, AND 5. The subjects should not participate in any other research protocols.

Exclusion Criteria:

1. Patients with pre-existing chronic facial pain not related to chronic rhinosinusitis.
2. Patients with pre-existing chronic pain of different etiology.
3. Patients taking prescription pain medications.
4. Patients taking antidepressant medications.
5. Patients taking over-the-counter pain medications within 48 hours of scheduled surgery.
6. Patients in whom oral opioid-containing analgesics would be contraindicated postoperatively.
7. Patients with a known or suspected genetic susceptibility to malignant hyperthermia, or known sensitivity to Desflurane or other halogenated agents.
8. Patients with the history of arrhythmias or significant coronary artery disease.
9. Patients with psychological disorders.
10. Patients who are unable to understand the questionnaires or the visual analogue scale (VAS) pain scores.
11. Patients with the history of substance or alcohol abuse.
12. Patients with compromised renal and liver function.
13. Patients with abnormal coagulation status or platelet count less than 100,000.
14. Pregnant patients.
15. Patients with an allergy to Bupivacaine, Lidocaine or Epinephrine.
16. Other patients that may be excluded by the investigator, based on medical history and physical examination

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2007-08; Primary Completion 2010-03 (Actual); Study Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David R. Drover, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

REFERENCES:
- [Result] Cho DY, Drover DR, Nekhendzy V, Butwick AJ, Collins J, Hwang PH. The effectiveness of preemptive sphenopalatine ganglion block on postoperative pain and functional outcomes after functional endoscopic sinus surgery. Int Forum Allergy Rhinol. 2011 May-Jun;1(3):212-8. doi: 10.1002/alr.20040. Epub 2011 Apr 13. PMID 22287376

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Stanford medical center
Pre-assignment Details: Having unilateral FESS
Groups:
- Group 1 - Bupivacaine Block: Active treatment group with application of bupivacaine block before FESS.
- Group 2 - Placebo Saline Block: This group proceeded as per teh active treatment group but with blinded use of saline in the block syringe before start of FESS.
Period: Overall Study
Arm/Group | Group 1 - Bupivacaine Block | Group 2 - Placebo Saline Block
Started | 29 | 27
Completed | 29 | 27
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Group 1 Bupivacaine: Active treatment group with application of bupivacaine block before FESS.
- Group 2 - Saline Placebo Group: Saline substituted in block, placebo treatment group with application of saline block before FESS.
- Total: Total of all reporting groups
Arm/Group | Group 1 Bupivacaine | Group 2 - Saline Placebo Group | Total
Number analyzed (Participants) | 29 | 27 | 56
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1 | 1 | 2
  Between 18 and 65 years | 26 | 21 | 47
  >=65 years | 2 | 5 | 7
Age, Continuous [Mean (Full Range); unit: years] | 49 [18 to 75] | 42 [18 to 67] | 45 [18 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 7 | 15
  Male | 21 | 20 | 41
Region of Enrollment [Number; unit: participants]
  United States | 29 | 27 | 56

OUTCOME MEASURES:

1. Primary Outcome: Postoperative Pain Assessed on Standard VAS Scale
Description: Post-operative quality of recovery and pain followed up to 1 month. Visual Analog Pain (VAS) was recorded by the patient on a 10-centimeter line to mark an estimated pain score that could be from zero (0) to ten (10). Zero would indicate no pain while a score of 10 would be the worse pain possible.
Time Frame: VAS Pain Score at 7 days
Population: Entire population of both groups.
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: VAS
Arm/Group | 1 - Bupivacaine Block | 2 - Placebo
Number analyzed (Participants) | 29 | 27
Number analyzed (VAS) | 29 | 27
units on a scale | 0.48 (0.23) | 1.12 (0.3)

2. Secondary Outcome: SNOT-20 Surgical Outcome Score
Description: This measures uses a 20 item surgical assessment tool to assess surgical field. This assessment score is the Sino-Nasal Outcome Test, SNOT-20. Patients were completed this validated sinus symptom questionnaire. The average magnitude score for the 20 items is calculated. Each item of the 20-question assessment is scored from 1 to 5 where 1 is less severe and 5 is a maximum as described by that particular symptom score. The final score is reported as a mean with a range of 0 (zero) to 5 (no units).
  ref. Otolaryngol Head Neck Surg, 126 (2002), pp. 41-47
Time Frame: 1-day
Population: Entire study population included.
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: Score
Arm/Group | Group 1 - Bupivacaine Block | Group 2 - Placebo Saline Block
Number analyzed (Participants) | 29 | 27
Number analyzed (Score) | 29 | 27
units on a scale | 1.76 (0.2) | 1.67 (0.2)

ADVERSE EVENTS:
Time Frame: From time of enrollment until the 30-day follow-up visit.
Groups:
- Group 1 - Bupicaine Block: Active treatment group with application of bupivacaine block before FESS.
- Group 2 - Saline Placebo Block: Placebo treatment group with application of saline block before FESS.
Arm/Group | Group 1 - Bupicaine Block | Group 2 - Saline Placebo Block
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/27
Other Adverse Events (participants affected / at risk) | 0/29 | 0/27

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No